CLINICAL TRIAL: NCT00753077
Title: Three Dimensional Morphology of Upper Respiratory Tract and Mandibular Position on Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, hospital, National Taiwan University Hospital
Other Study IDs: 200804052R
Record Dates: First submitted 2008-09-14; First posted 2008-09-16 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Oral appliances, which can maintain patients' jaw forwards during sleep, become more popular in treating obstructive sleep apnea (OSA). However, the exact mechanism of mandible forward on upper airway is not completely known. In this study we will use both static and dynamic MRI to study the 3D morphological changes and dynamic behavior of the upper respiratory tract at different mandible posits. Because in asian society non-obese OSA patients are not uncommonly seen, in this study we focus only on non-obese severe OSA patients.

DETAILED DESCRIPTION:
The aim of this study is to analyze upper airway morphology changes and dynamic movement at different sections affected by mandible position by using dynamic and static magnet resonance imaging technique. The study also discusses the formation mechanism of obstructive sleep apnea syndromes and function mechanism of the oral appliance, as well as the evaluation of the clinical results of the oral appliance on non-obese male patients with severe obstructive sleep apnea in Taiwan.

10 non-obese (BMI<25) severe OSA (AHI>30) male patients between the age of 20 to 60 and 10 gender, BMI and age matched control (AHI<5) were recruited for this study. Nine bite index were made for the different mandible positions of the subjects.

Upper airway was imaged by using static and dynamic MRI of each subject wearing the bite index while lying on the MRI scanning table. This study also measures the circumference and takes the lateral cephalometric imaging of each subject. Oral appliances were made and fitted for the experimental group subjects, who wore them for three months, after which they transferred to the Sleep Center and underwent PSG examination to evaluate therapeutic effects of the appliances.

ELIGIBILITY:
Inclusion Criteria:

* Severe obstructive sleep apnea (AHI>=30/hr) age, sex, BMI match control subject

Exclusion Criteria:

* Patients were excluded when:

  * (1) refused to participate in this study,
  * (2) had severe obstructive pulmonary disease or active neurological events,
  * (3) enrolled in other studies at the same time

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients referred from sleep center
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, National Taiwan University, Taipei, Taiwan